CLINICAL TRIAL: NCT03031691
Title: A Phase 1b Dose Escalation Study of the Safety and Pharmacodynamics of Brontictuzumab in Combination With Chemotherapy for Subjects With Previously Treated Metastatic Colorectal Cancer
Brief Title: A Study of Brontictuzumab With Chemotherapy for Subjects With Previously Treated Metastatic Colorectal Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: OncoMed Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Organization: Mereo BioPharma (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 52M51-003
Record Dates: First submitted 2017-01-13; First posted 2017-01-25 (Estimated); Last update posted 2020-08-11 (Actual); Status verified 2020-08

CONDITIONS: Metastatic Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — trifluridine tipiracil drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Brontictuzumab and trifluridine/tipiracil (Experimental): Brontictuzumab will be administered per protocol and trifluridine/tipiracil per label.
  Interventions: Drug: brontictuzumab; Drug: trifluridine/tipiracil

INTERVENTIONS:
Drug: brontictuzumab — starting dose of 1.5mg/kg administered intravenously (IV)
  Other Names: OMP-52M51
Drug: trifluridine/tipiracil

SUMMARY:
A Phase 1b Dose Escalation Study of the Safety and Pharmacodynamics of Brontictuzumab in Combination with Chemotherapy for Subjects with Previously Treated Metastatic Colorectal Cancer.

DETAILED DESCRIPTION:
This is a phase 1b dose escalation study of the safety and pharmacodynamics of brontictuzumab in combination with chemotherapy for subjects with previously treated metastatic colorectal cancer. This study consists of a screening period, a treatment period and a post-treatment follow up period in which patients will be followed for survival for up to 24 months. Patients will be enrolled in two stages: a dose-escalation stage and an expansion phase.

Approximately 34 patients will be enrolled in this study at approximately 5 study centers in the United States.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed metastatic colorectal cancer (mCRC) previously treated with fluoropyrimidine-, oxaliplatin- and irinotecan-based chemotherapy, an anti-VEGF biological therapy, and if KRAS wild-type, an anti-EGFR therapy
* ECOG performance status 0 or 1

Exclusion Criteria:

* Prior treatment with gamma secretase inhibitors or other Notch 1 inhibitors
* Subjects with known active HIV infection. Subjects with HIV that are under a stable anti-retroviral regimen and have no evidence of immune deficiency (normal CD4 counts), undetectable viral load, and no HIV-related infections are eligible
* Subjects with uncontrolled diarrhea <30 days prior to first administration of study drug
* Subjects with any history of or current clinically significant gastrointestinal disease including, but not limited to:

  * Inflammatory bowel disease (including ulcerative colitis and Crohn's disease)
  * Active peptic ulcer disease
  * Known intraluminal metastatic lesion(s) with risk of bleeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2017-01; Primary Completion 2017-05 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with adverse events | up to approximately 2 years
Percentage of patients with dose limiting toxicities | 28 days
Percentage of patients with anti-brontictuzumab antibodies | up to approximately 2 years

SECONDARY OUTCOMES:
Objective Response according to Response Evaluation Criteria in Solid Tumors (RECIST 1.1) | approximately 2 years
Progression-free survival according to Response Evaluation Criteria in Solid Tumors (RECIST 1.1 | approximately 2 years
Changes in number of circulating tumor cells | approximately 2 years
Overall survival | approximately 2 years

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Denver, Denver, Colorado
  - Miami, Miami, Florida
  - Sarasota, Sarasota, Florida
  - Charleston, Charleston, South Carolina
  - Nashville, Nashville, Tennessee